CLINICAL TRIAL: NCT01908582
Title: Effect of Rifampin on the Pharmacokinetics of Evacetrapib in Healthy Subjects
Brief Title: A Study of Evacetrapib and Rifampin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14636; I1V-MC-EIAZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (Experimental): Period 1:
  130 milligram (mg) evacetrapib administered orally, once on Day 1
  Interventions: Drug: Evacetrapib
- Evacetrapib + Rifampin (Experimental): Period 2:
  Rifampin: 600 mg administered orally, once daily (QD) for 14 days (Days 9 to 22)
  Evacetrapib: 130 mg administered orally once on Day 16
  Interventions: Drug: Evacetrapib; Drug: Rifampin

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
Drug: Rifampin — Administered orally
  Arms: Evacetrapib + Rifampin

SUMMARY:
The main purpose of this study is to determine how much evacetrapib gets into the blood stream and how long it takes the body to get rid of it when given with rifampin. The safety and tolerability of the two drugs, given together, will also be evaluated. The study will also look at blood cholesterol levels and levels of a hormone called cortisol before and after taking rifampin. Information about any side effects that may occur will also be collected.

For each participant, this study will include 2 periods in fixed order. The study will last approximately 29 days.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males and females (of non child-bearing potential)
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Have known allergies to evacetrapib, rifampin, related compounds or any components of either formulation, or history of significant allergic disease as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Period 1:
  Evacetrapib 130 milligrams (mg) administered orally as a single dose on Day 1
  Period 2:
  Rifampin 600 mg administered orally once daily (QD) of Days 9 to 22 Evacetrapib 130 mg administered orally as a single dose on Day 16
Period: Period 1
Arm/Group | All Participants
Started | 26
Received at Least One Dose of Study Drug | 26
Completed | 26
Not Completed | 0
Period: Period 2
Arm/Group | All Participants
Started | 26
Completed | 24
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Participants: Period 1:
  Evacetrapib 130 mg administered orally as a single dose on Day 1
  Period 2:
  Rifampin 600 mg administered orally QD of Days 9 to 22 Evacetrapib 130 mg administered orally as a single dose on Day 16
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Evacetrapib
Time Frame: Day 1 and Day 16, predose of evacetrapib and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of rifampin or evacetrapib and had evaluable evacetrapib concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Evacetrapib: Period 1:
  Evacetrapib 130 mg administered orally as a single dose on Day 1
- Evacetrapib + Rifampin: Period 2:
  Rifampin 600 mg administered orally, QD on Days 9 to 22 (14 consecutive days)
  Evacetrapib 130 mg administered orally as a single dose on Day 16
Arm/Group | Evacetrapib | Evacetrapib + Rifampin
Number analyzed (Participants) | 25 | 25
nanograms per milliliter (ng/mL) | 599 (64) | 269 (55)

2. Primary Outcome: Pharmacokinetics (PK): Time of Maximum Observed Drug Concentration (Tmax) of Evacetrapib
Time Frame: Day 1 and Day 16, predose of evacetrapib and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Evacetrapib | Evacetrapib + Rifampin
Number analyzed (Participants) | 25 | 25
hours | 2.00 [2.00 to 4.00] | 2.00 [1.00 to 6.00]

3. Primary Outcome: Pharmacokinetics, Area Under the Plasma Concentration-Time Curve From Time 0 Hour (h) to Infinity (AUC0-∞) of Evacetrapib
Time Frame: Day 1 and Day 16, predose of evacetrapib and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All participants who received at least 1 dose of evacetrapib and have evaluable evacetrapib concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hours per milliliter
Arm/Group | Evacetrapib | Evacetrapib + Rifampin
Number analyzed (Participants) | 25 | 24
nanograms * hours per milliliter | 9810 (47) | 2070 (42)

ADVERSE EVENTS:
Groups:
- Rifampin: Period 2:
  600 mg rifampin administered orally as a single dose QD on Days 9 through 15.
- Evacetrapib + Rifampin: Period 2:
  Rifampin 600 mg administered orally, QD on Days 16 to 22
  Evacetrapib 130 mg administered orally as a single dose on Day 16
Arm/Group | Evacetrapib | Rifampin | Evacetrapib + Rifampin
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 26/26 | 5/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (N=26) | Rifampin (N=26) | Evacetrapib + Rifampin (N=26)
Vessel puncture site pain (General disorders) | 1 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3)
Chromaturia (Renal and urinary disorders) | 0 (0) | 26 (26) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days